CLINICAL TRIAL: NCT06094569
Title: Medical Imaging Screening for Posterior-circulation Ischemic Stroke：a Multicentre,Imaging-based,Prospective Cohort Study
Brief Title: Medical Imaging Screening for Posterior-circulation Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Other Study IDs: TJHH-2023-wm14
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Endovascular Thrombectomy
Keywords: select patients; endovascular thrombectomy; magnetic resonance imaging; diffusion weighted imaging; Vertebrobasilar artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular therapy: Timely thrombectomy for acute ischemic stroke patients with large vessel occlusion by either stent retriever, thrombus aspiration, others, or combination methods.
  Interventions: Procedure: Endovascular Therapy
- Best medical management: Patients enrolled in this group received the best medical management.

INTERVENTIONS:
Procedure: Endovascular Therapy — Endovascular therapy, as an adjunct to standard stroke therapy, may be beneficial for a very select population of patients who present with an acute ischemic stroke and have a proven large, proximal occlusion on imaging. Endovascular therapy includes any one or more of the following: Intra-arterial thrombolytic therapy, aspiration, stent retrieval, or a combination of multiple mechanical devices
  Groups: Endovascular therapy

SUMMARY:
Patients with ischemic stroke in the posterior circulation continue to have high rates of mortality and disability, even with aggressive treatment. We wanted to evaluate preoperative imaging to screen patients with a good prognosis from mechanical embolization. We assess the degree of ischemia by defining the pons-midbrain-medulla index (PMMI) and correlate the preoperative PMMI with the clinical prognosis of postoperative patients to verify the validity of PMMI in predicting the clinical prognosis of patients with embolization.

DETAILED DESCRIPTION:
* The ENDOSTROKE registry (Endovascular Stroke T reatment Registry), the use of MRI before EVT was associated with significantly better clinical outcomes as compared to CT.
* The purpose of the study will sift patients with posterior circulation ischemia stroke who will get better outcome by Mechanical Thrombectomy by neuroimaging.Specifically, the following assumption will be evaluated: the modified pons-midbrain index in magnetic resonance imaging can predict the clinical outcome of patients with basilar artery thrombosis 90 days after surgery, and can guide whether patients will undergo mechanical thrombectomy later.
* Pons-midbrain-medulla index (PMMI) : We divide pons-midbrain-medulla into the left and right sides by the median line of the brainstem,so we will evaluate ischemia of these six layers which are endowed different score according to the degree of ischemia. Instead of the previous pons-midbrain index (PMI), we select the image layer that shows the largest infarct size among the six parts.Then,we add up six scores that is patient's PMMI. Scoring criteria: At the layer of displaying the maximum infarct size, 2 points are scored if the infarct size exceeds 50% of the total area, 1 point is scored if the infarct size is less than 50% of the total area, and 0 points are scored if there is no infarct.Finally, PMMI values range from 0 to 12 points.
* The investigators conduct a multicenter, prospective cohort study.Preoperative images of patients are evaluated by different groups of imaging physicians to describe the association between preoperative PMMI and clinical prognosis in patients with posterior circulation stroke and to verify its validity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient admitted from Jun. 1st 2019 to Jan. 1st 2029;
2. Patients with acute ischemic stroke recently；
3. Symptoms persisted at admission, and MRI (including DWI) confirmed acute ischemic vertebrobasilar artery occlusion in the posterior circulation:（single right or left intracranial branch of vertebral artery occlusion ; single basilar occlusion ; both two vertebral arterys and basilar artery）；

Exclusion Criteria:

1.Patiens can not meet the MRI examination conditions(with absolute and relative contraindications).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All acute ischemic strvoke patients with vertebrobasilar artery occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified ranking scale (mRS) at 90 days | 90 days
  A 0-6 scale running from perfect health without symptoms to death.

SECONDARY OUTCOMES:
Mortality within 90 days | 90 days
  mortality of any causes.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) scores at 90 days | 90 days
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Occurrence of periprocedural complications | 90 days
  Periprocedural complications include any intracranial hemorrhage, cerebral edema, brain herniation and pneumonia.
pc-ASPECT (posterior circulation Alberta Stroke Program Early CT score) | 0 days
  pc-ASPECTS is a 10-point quantitative topographic CT scan score used in patients with posterior circulation stroke.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The Sencond Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Beijing University Binhai Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided